CLINICAL TRIAL: NCT05813613
Title: Role of Artificial Intelligence in Predicting Muscle Fatigue Using Virtual Reality Training In Healthy And Post COVID19 Subjects
Brief Title: Role of Artificial Intelligence in Predicting Muscle Fatigue Using Virtual Reality Training
Status: Completed | Type: Observational
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Rami Abbas, Associate. Prof. Rami Abbas, Beirut Arab University
Other Study IDs: AI in Prediciting Fatigue
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Fatigue
Keywords: Electromyography; Fatigue; Squats; Borg scale; Musculoskeletal disorders
MeSH Terms: conditions — Fatigue; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Group: * Will perform squatting exercise while reporting subjective muscle fatigue levels periodically, until maximal subjective fatigue is reached
  * Will have sEMG for vastus lateralis and rectus femoris, chest expansion, goniometry for the knee recording using the Biopac.
  Interventions: Other: Squatting with the aid of Kynapsis Virtual Training apparatus.
- Post Covid-19 Group: * Will perform squatting exercise while reporting subjective muscle fatigue levels periodically, until maximal subjective fatigue is reached
  * Will have sEMG for vastus lateralis and rectus femoris, chest expansion, goniometry for the knee recording using the Biopac.
  Interventions: Other: Squatting with the aid of Kynapsis Virtual Training apparatus.

INTERVENTIONS:
Other: Squatting with the aid of Kynapsis Virtual Training apparatus. — Squatting exercise was performed using a virtual reality (VR) machine (kynapsis) for guidance in both groups. Squats were performed while the hands were kept in front of the bodies and the knees flexed to 90 degrees following a rhythm of two seconds for descent, two second ascent mimicking the movement done on the VR machine.

SUMMARY:
The goal of this observational predicted study is to predict muscle fatigue using a specific AI algorithm in healthy vs post Covid-19 infected individuals. The main question it aims to answer is:

Can Artificial Intelligence be used as a reliable source of predicting localized muscle fatigue in healthy vs post Covid-19 infected individuals?

Participants will be divided into two groups: A healthy group and a post Covid-19 group.

* Each group will undergo a familiarization process before the start of the exercises.
* Then, each group will perform squatting exercises guided by the kynpasis virtual reality apparatus.
* sEMG for the vastus lateralis and rectus femories, chest expansion, and goniometric measurements of the knee will be taken during different reported fatigue levels using the Biopac system.
* Groups will continue squatting while recording their subjective fatigue levels using the Borg scale.
* Data will then be run through machine learning processes to produce an AI algorithm capable of predicting isolated muscle fatigue.

DETAILED DESCRIPTION:
Participants were divided into two groups, one consisting of healthy individuals and another consisting of Covid-19 subjects. Both groups received a familiarization training for the exercise to be performed with 15 minutes of rest afterwards, before the start of the data collection.

Squatting exercise was performed using a virtual reality (VR) machine (kynapsis) for guidance in both groups. Squats were performed while the hands were kept in front of the bodies and the knees flexed to 90 degrees following a rhythm of two seconds for descent, two second ascent mimicking the movement done on the VR machine.

Additional variables were considered, including chest expansion, and the range of motion using an electric goniometer, all being measured and recorded using the Biopac (BIOPAC Systems, Inc., Santa Barbara, CA) that, according to evidence, possess a high-pass frequency filter and bipolar electrode system.

The muscles tested are the 3 heads of the QF muscle RF, VM, and VL. Their areas were cleaned using alcohol and shaved to reduce resistance of electrodes. Three disposable sEMG surface electrodes were placed, two of them on the muscle belly with 2.5cm distance between them, and one control electrode placed on the agonist side, the participant was asked to extend their knee and flex it against resistance to locate the lateral and medial vasti. sEMG electrodes were placed on the subdivisions of the QF muscle during the exercise. The extracted data is then run through an AI algorithm that will analyze and predict muscle fatigue.

The Borg (C-10) scale was explained to the participants and was present in front of them while performing the exercise as an outcome measure to assess the subjective muscle fatigue that once reached will end the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Non-athletic healthy individuals.
* Avoided intense activities in the past 3 days.
* Confirmed positive PCR test done within an interval of 1 year for Covid-19 group subjects.

Exclusion Criteria:

* Being old age geriatrics (more than 50 years old).
* Having any respiratory, cardiac, renal, neuromuscular, orthopedic, and musculoskeletal disorders.
* Smokers and some medicinal drug users must be taken into consideration because it affects the performance and increases the fatigue levels.
* Subjects not meeting any of the inclusion criteria.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of two groups.
  * Non-athletic healthy individuals that did not perform any intense activities for the past 3 days and had not contacted Covid-19 previously.
  * Non-athletic healthy individuals that did not perform any intense activities for the past 3 days but have a confirmed positive PCR test done within a 1 year interval.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Surface electromyography | During the squatting exercise.
  non-invasive technique where electrodes were placed on the vastus lateralis and rectus femoris heads of the quadriceps femoris muscle, assessing it's myoelectric output. Their areas were cleaned using alcohol and shaved to reduce resistance of electrodes. Three disposable sEMG surface electrodes were placed, two of them on the muscle belly with 2.5cm distance between them, and one control electrode placed on the agonist side, the participant was asked to extend their knee and flex it against resistance to locate the lateral and medial vasti. sEMG electrodes were placed on the subdivisions of the QF muscle during the exercise. The extracted data is then run through an AI algorithm that will analyze and predict muscle fatigue.
The Borg Rating of Perceived Exertion (RPE) scale | During the squatting exercise.
  A tool for measuring an individual's effort and exertion, breathlessness and fatigue during physical work and so is highly relevant for occupational health and safety practice. It ranges from 6 as a minimum to 20 as a maximum with 6 signifying no exertion and 20 signifying extreme maximal exertion

SECONDARY OUTCOMES:
Chest Expansion. | During the squatting exercise.
  Using a respiration transducer wrapped around the subject's chest using a velcro strap that transmits expansion data to the main receiver module of the Biopac, that will be recorded on the computer.
Range of motion. | During the squatting exercise.
  Using an electric goniometer wired on the subject's knee that will transmit signals of range of motion to the receiver module of the Biopac that will be recorded on the computer.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad ElMelhat, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wan JJ, Qin Z, Wang PY, Sun Y, Liu X. Muscle fatigue: general understanding and treatment. Exp Mol Med. 2017 Oct 6;49(10):e384. doi: 10.1038/emm.2017.194. PMID 28983090
- [Background] A narrative review of immersive virtual reality's ergonomics and risks at the workplace: cybersickness, visual fatigue, muscular fatigue, acute stress, and mental overload Souchet, A.D., Lourdeaux, D., Pagani, A. et al. A narrative review of immersive virtual reality's ergonomics and risks at the workplace: cybersickness, visual fatigue, muscular fatigue, acute stress, and mental overload. Virtual Reality (2022). https://doi.org/10.1007/s10055-022-00672-0
- [Background] Donatelli, R.A. (2007) Sports-specific rehabilitation. St. Louis, MO: Churchill Livingstone.
- [Background] Hall, J. E., & Hall, M. E. (2020). Guyton and Hall textbook of medical physiology e-Book. Elsevier Health Sciences.
- [Background] Paneroni M, Simonelli C, Saleri M, Bertacchini L, Venturelli M, Troosters T, Ambrosino N, Vitacca M. Muscle Strength and Physical Performance in Patients Without Previous Disabilities Recovering From COVID-19 Pneumonia. Am J Phys Med Rehabil. 2021 Feb 1;100(2):105-109. doi: 10.1097/PHM.0000000000001641. PMID 33181531
- [Background] Schoenfeld BJ. Squatting kinematics and kinetics and their application to exercise performance. J Strength Cond Res. 2010 Dec;24(12):3497-506. doi: 10.1519/JSC.0b013e3181bac2d7. PMID 20182386
- [Background] Kubo K, Ikebukuro T, Yata H. Effects of squat training with different depths on lower limb muscle volumes. Eur J Appl Physiol. 2019 Sep;119(9):1933-1942. doi: 10.1007/s00421-019-04181-y. Epub 2019 Jun 22. PMID 31230110
- [Background] Davenport T, Kalakota R. The potential for artificial intelligence in healthcare. Future Healthc J. 2019 Jun;6(2):94-98. doi: 10.7861/futurehosp.6-2-94. PMID 31363513
- [Background] Tack C. Artificial intelligence and machine learning | applications in musculoskeletal physiotherapy. Musculoskelet Sci Pract. 2019 Feb;39:164-169. doi: 10.1016/j.msksp.2018.11.012. Epub 2018 Nov 23. PMID 30502096
- [Background] Luna A, Casertano L, Timmerberg J, O'Neil M, Machowsky J, Leu CS, Lin J, Fang Z, Douglas W, Agrawal S. Artificial intelligence application versus physical therapist for squat evaluation: a randomized controlled trial. Sci Rep. 2021 Sep 13;11(1):18109. doi: 10.1038/s41598-021-97343-y. PMID 34518568
- [Background] Alsobhi M, Khan F, Chevidikunnan MF, Basuodan R, Shawli L, Neamatallah Z. Physical Therapists' Knowledge and Attitudes Regarding Artificial Intelligence Applications in Health Care and Rehabilitation: Cross-sectional Study. J Med Internet Res. 2022 Oct 20;24(10):e39565. doi: 10.2196/39565. PMID 36264614
- [Background] Qian J, McDonough DJ, Gao Z. The Effectiveness of Virtual Reality Exercise on Individual's Physiological, Psychological and Rehabilitative Outcomes: A Systematic Review. Int J Environ Res Public Health. 2020 Jun 10;17(11):4133. doi: 10.3390/ijerph17114133. PMID 32531906
- [Background] Sun J, Liu G, Sun Y, Lin K, Zhou Z, Cai J. Application of Surface Electromyography in Exercise Fatigue: A Review. Front Syst Neurosci. 2022 Aug 11;16:893275. doi: 10.3389/fnsys.2022.893275. eCollection 2022. PMID 36032326
- [Background] Al-Mulla MR, Sepulveda F, Colley M. An autonomous wearable system for predicting and detecting localised muscle fatigue. Sensors (Basel). 2011;11(2):1542-57. doi: 10.3390/s110201542. Epub 2011 Jan 27. PMID 22319367
- [Background] Calder KM, Stashuk DW, McLean L. Physiological characteristics of motor units in the brachioradialis muscle across fatiguing low-level isometric contractions. J Electromyogr Kinesiol. 2008 Feb;18(1):2-15. doi: 10.1016/j.jelekin.2006.08.012. Epub 2006 Nov 20. PMID 17113787
- [Background] Torvik, G. I., Triantaphyllou, E., Liao, T., & Waly, S. (1999, March). Predicting muscle fatigue via electromyography: A comparative study. In Proceedings of the 25th International Conference on Computers and Industrial Engineering (pp. 277-280)
- [Background] Caesaria, A. P., Endro Yulianto, Luthfiyah, S., Triwiyanto, T., & Rizal, A. (2023). Effect of Muscle Fatigue on EMG Signal and Maximum Heart Rate for Pre and Post Physical Activity. Journal of Electronics, Electromedical Engineering, and Medical Informatics, 5(1), 39-45. https://doi.org/10.35882/jeeemi.v5i1.278
- [Background] Ahmad I, Kim JY. Assessment of Whole Body and Local Muscle Fatigue Using Electromyography and a Perceived Exertion Scale for Squat Lifting. Int J Environ Res Public Health. 2018 Apr 18;15(4):784. doi: 10.3390/ijerph15040784. PMID 29670002
- [Background] Disser NP, De Micheli AJ, Schonk MM, Konnaris MA, Piacentini AN, Edon DL, Toresdahl BG, Rodeo SA, Casey EK, Mendias CL. Musculoskeletal Consequences of COVID-19. J Bone Joint Surg Am. 2020 Jul 15;102(14):1197-1204. doi: 10.2106/JBJS.20.00847. PMID 32675661
- [Background] Dos Santos PK, Sigoli E, Braganca LJG, Cornachione AS. The Musculoskeletal Involvement After Mild to Moderate COVID-19 Infection. Front Physiol. 2022 Mar 18;13:813924. doi: 10.3389/fphys.2022.813924. eCollection 2022. PMID 35492595
- [Background] Diem L, Fregolente-Gomes L, Warncke JD, Hammer H, Friedli C, Kamber N, Jung S, Bigi S, Funke-Chambour M, Chan A, Bassetti CL, Salmen A, Hoepner R. Fatigue in Post-COVID-19 Syndrome: Clinical Phenomenology, Comorbidities and Association With Initial Course of COVID-19. J Cent Nerv Syst Dis. 2022 May 24;14:11795735221102727. doi: 10.1177/11795735221102727. eCollection 2022. PMID 35633835
- [Background] Ducrocq GP, Blain GM. Relationship between neuromuscular fatigue, muscle activation and the work done above the critical power during severe-intensity exercise. Exp Physiol. 2022 Apr;107(4):312-325. doi: 10.1113/EP090043. Epub 2022 Mar 4. PMID 35137992
- [Background] Joli J, Buck P, Zipfel S, Stengel A. Post-COVID-19 fatigue: A systematic review. Front Psychiatry. 2022 Aug 11;13:947973. doi: 10.3389/fpsyt.2022.947973. eCollection 2022. PMID 36032234
- [Background] Faulkner JA, Larkin LM, Claflin DR, Brooks SV. Age-related changes in the structure and function of skeletal muscles. Clin Exp Pharmacol Physiol. 2007 Nov;34(11):1091-6. doi: 10.1111/j.1440-1681.2007.04752.x. PMID 17880359